CLINICAL TRIAL: NCT02005016
Title: Dosage and Predictors of Naming Treatment Response in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O0832-R; 1I01RX000832-01A2 (NIH)
Record Dates: First submitted 2013-11-14; First posted 2013-12-09 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Language Therapy; Acquired Language Disorders; Semantics; Stroke
MeSH Terms: conditions — Aphasia; Stroke; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All study participants will be assigned to this arm of this single-arm study. Participants will receive intensive behavioral therapy intended to improve their naming (word production) ability.
  Interventions: Behavioral: Naming therapy

INTERVENTIONS:
Behavioral: Naming therapy — Participants will receive behavioral therapy which is designed to stimulate semantic (meaning) representations which are required for successful naming (word production). Therapy will be administered for 4 weeks on an intensive schedule (5 days a week, approximately 4.5 hours per day).
  Other Names: Semantic feature analysis

SUMMARY:
This study examines aphasia treatment response among Veterans and non-Veterans living with aphasia. It seeks to identify cognitive and neural factors which are predictive of positive response to treatment targeting naming impairments in aphasia. It also examines the dose-response relationship for naming treatment. More broadly, it seeks to determine who aphasia therapy works best for, and how much aphasia therapy is sufficient to achieve positive treatment response.

DETAILED DESCRIPTION:
Language and communicative impairments following stroke (aphasia) affect more than 30% of stroke survivors, with an incidence of over 180,000 new cases annually. The consequences of aphasia are far reaching and can affect psychosocial adjustment, family role participation, vocational opportunities, and the ability to function independently in society. Recent estimates suggest that VHA outpatient clinics see 2000 new cases of aphasia each year, meaning that approximately 20,000 enrolled VHA patients and 100,000 United States Veterans are currently living with the condition. In response to this need, the VA Pittsburgh Healthcare System Geriatric Research, Education, and Clinical Center (GRECC) initiated the Program for Intensive Residential Aphasia Treatment and Education (PIRATE) in January 2009. PIRATE is a clinical demonstration project that provides approximately 100 hours of cognitive-linguistically oriented aphasia treatment to community dwelling Veterans over a 4-week period. PIRATE currently serves 18 Veterans per year in bi-monthly sessions. Resource limitations associated with PIRATE and aphasia treatment in general require that treatments be offered in the most cost-effective doses to those Veterans most likely to benefit from them.

This treatment-effectiveness research study addresses these issues by examining the dose-response relationship for semantically-oriented naming treatment, and identifying cognitive, psycholinguistic and neuroanatomical predictors of treatment success. Study participants (n=60, over a 4-year period) will be recruited nationwide from Veterans enrolled in PIRATE. They will have their naming performance measured prior to PIRATE entry, during each week of treatment, and at program exit/follow-up. A battery of cognitive measures and structural magnetic resonance images of their brains will also be collected prior to treatment. Participants' performance on trained and untrained lexical items and a standardized measure of naming performance will be compared across time intervals to specify the therapy amounts for which maximum treatment benefits are achieved. Their treatment outcomes will also be correlated with specific cognitive test scores and the location and extent of their brain lesions to identify cognitive and neurological markers predictive of positive treatment response. Treatment response will also be compared across participants with different psycholinguistic profiles, to determine which groups of patients show greatest benefit from semantically-oriented naming treatment.

This study should provide answers to two interlocking questions: for whom is aphasia therapy most effective, and how much of it is needed to optimize treatment outcomes. These answers have the potential to set transformative new standards for how aphasia treatment is delivered within VHA and to stroke survivors with aphasia more broadly.

ELIGIBILITY:
Inclusion Criteria:

* All study participants will be community-dwelling adults with aphasia.
* Both Veterans and non-Veterans who are able to arrange daily transportation to and from the campus of the VA Pittsburgh Healthcare System (VAPHS), and who do not require housing, may be eligible to be study participants.
* In addition, Veterans who are accepted into the Program for Intensive Residential Aphasia Treatment and Education (PIRATE) of VAPHS may be eligible to participate.

  * PIRATE participants are Veterans who are referred nationally to VAPHS.
  * Aphasia diagnosis is provided by the referring medical provider, based on performance on standardized aphasia-assessment measures, and will be verified by PIRATE staff prior to enrollment. Diagnosis will be based on clinical impression and performance on the Comprehensive Aphasia Test (CAT).

Study participants must also meet the following inclusion criteria:

* 18 years of age or older
* Eligible for participation in the standard PIRATE program
* Aphasia due to unilateral left hemisphere stroke equal to or more than 6 months post onset
* Overall CAT mean language modality t-score of less than or equal to 70
* CAT naming modality t-score greater than or equal to 40
* No progressive neurological disease or prior central nervous system injury/disorder
* No severe motor speech disorders (apraxia and/or dysarthria)
* Learned English as a first language
* Investigators able to construct lists of sufficient treatment targets and generalization probes based on performance on naming assessments

Exclusion Criteria:

Since all study candidates must be present on the VAPHS campus for treatment, and must undergo intensive speech-language therapy (up to 5 hours per day for 4 weeks), the following exclusionary criteria apply to all participants:

* Inability to carry out activities of daily living necessary for self-care during the time they are present on the VAPHS campus
* Lack of physical independence which would interfere with their ability to be present on the VAPHS campus
* History of progressive neurological disease
* History of drug or alcohol dependence that is not currently stable/medically managed
* Inability to tolerate intensive treatment as determined by previous therapy experiences and tolerance of the intensive initial evaluation (2 days of testing)

In addition, participants who are enrolling in the study through the PIRATE program have the following exclusion criteria apply:

* Inability to carry out activities of daily living necessary for self-care as determined by an occupational therapy assessment prior to program entry
* Lack of physical independence
* History of significant mood or behavioral disorder that is not currently stable/medically managed
* History of progressive neurological disease
* History of drug or alcohol dependence that is not currently stable/medically managed
* Inability to tolerate intensive treatment as determined by previous therapy experiences and tolerance of the intensive initial evaluation (2 days of testing)
* Medical conditions which would preclude independent living as determined by the medical assessment provided by a VAPHS physician prior to program entry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Dickey, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Dosage and Predictors of Naming Treatment Response in Aphasia — http://www.pittsburgh.va.gov/PIRATE/

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Therapy: All study participants will be assigned to this arm of this single-arm study. Participants will receive intensive behavioral therapy intended to improve their naming (word production) ability.
  Naming therapy: Participants will receive behavioral therapy which is designed to stimulate semantic (meaning) representations which are required for successful naming (word production). Therapy will be administered for 4 weeks on an intensive schedule (5 days a week, approximately 4.5 hours per day).
Period: Overall Study
Arm/Group | Behavioral Therapy
Started | 46
Completed | 44
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants] — Population: Two enrolled participants did not complete the protocol.
  Participants
    number analyzed (Participants) | 44
    <=18 years | 0
    Between 18 and 65 years | 22
    >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.56 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 39
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46
Philadelphia Naming Test [Mean (Standard Deviation); unit: units on a scale] — The Philadelphia Naming Test (PNT) is a performance-based measure commonly used to assess naming (word production) ability among adults with aphasia. Participants are shown 175 pictures of common objects and asked to name each stimulus item within 30 seconds. Score range is from 0 to 175 (number out of 175 items that were correctly named), with higher scores representing better performance. Baseline PNT measures indicate pre-treatment naming (word production) ability.
  units on a scale | 111.96 (39.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Philadelphia Naming Test Score
Description: The Philadelphia Naming Test is a performance-based measure commonly used to assess naming (word production) ability among adults with aphasia. Participants are shown 175 pictures of common objects and asked to name each stimulus item within 30 seconds. Score range is from 0 to 175 (number out of 175 items that were correctly named), with higher scores representing better performance. Change in PNT score from entry to exit is the primary study outcome. Mean PNT change score measures treatment-related changes in naming ability.
Time Frame: Baseline (at study entry) to the day after completion of intervention (after 4 weeks of behavioral therapy).
Population: The PNT was administered at two timepoints for the majority of the sample (32/44). The initial 12 participants received the PNT at study entry and abbreviated forms of the assessment during the protocol and at study exit. These abbreviated forms were found not to be reliable, so the full PNT was administered to remaining participants at exit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 32
score on a scale | 5.91 (1.84)
Statistical Analysis 1: Comparison: Behavioral Therapy; Test type: Other — This was a single-group study. A t-test was administered comparing pre- and post-treatment PNT scores (range: 1-175; higher scores are better); p < 0.005, t-test, 1 sided

2. Secondary Outcome: Change From Baseline on Comprehensive Aphasia Test Modality Mean T-Score
Description: The Comprehensive Aphasia Test (CAT) is a performance-based measure of language processing across multiple language domains commonly used to assess language-processing ability among adults with aphasia. The CAT Modality Mean T-Score represents an measurement of overall language-processing ability (aphasia severity). Scores are on a T-score scale (mean score 50, 2 SD range from 30 to 70), with higher scores representing better performance. Change in CAT score from entry to exit (secondary outcome) measures treatment-related changes in overall aphasia severity.
Time Frame: Baseline (at study entry) to the day after completion of intervention (after 4 weeks of behavioral therapy).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 44
units on a scale | 0.80 (0.17)
Statistical Analysis 1: Comparison: Behavioral Therapy; Test type: Other — This was a single-group study. A t-test was administered comparing pre- and post-treatment CAT modality mean T-scores (range: 30-70, mean: 50; higher scores are better); p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant were collected over the period from baseline (study entry) to the day after completion of intervention (after 4 weeks of behavioral therapy).
Arm/Group | Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

LIMITATIONS AND CAVEATS:
The full PNT (primary outcome measure) was administered at entry and exit for a subset of the sample (32/44). 12 participants received the full PNT at entry but received abbreviated forms at exit; these forms were found not to be reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT02005016/Prot_SAP_000.pdf